CLINICAL TRIAL: NCT03825653
Title: Biomechanical Aligment of Lower Limb as a Predictor for Stress Urinary Incontinence in Postmenopasual Women
Brief Title: Biomechanical Aligment of Lower Limb as a Predictor for Stress Urinary Incontinence in Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, lecturer of biomechanics, Cairo University
Other Study IDs: P.T.REC/012/001885
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-12

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; pelvic tilt; ankle position
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: This study will be carried out on three hundred postmenopausal.They will be selected from gynecological outpatient clinic of (Oum El Masryn Hospital).
  their age will range from 60-70 years.Their BMI will not exceed 30 kg/m2. They are complaining from stress urinary incontinence.

SUMMARY:
This study will be conducted to assess biomechanical alignment of lower limb as a predictor for the stress urinary incontinence in the postmenopausal women. 300 postmenopausual women will be selected suffering from stress unrinary incontinence . Their age ranges from 60 to 70 years old. Their BMI is not exceeding 30 kg/m2.

DETAILED DESCRIPTION:
in this study 300 postmenopausual women will be selected suffering from stress unrinary incontinence. Their age ranges from 60 to 70 years old. Their BMI is not exceeding 30 kg/m2. different methods of assessment will be used as : Data recording sheet, Weight-Height scale, Goniometer ,x ray radiography ,Transabdominal ultrasound and Perineal ultrasound. Data recording sheet: It will be used to record data of each woman before starting this study. Weight-Height scale: It will be used to measure weight and height of each woman before starting this study. Goniometer: it will be used to document the initial and the subsequent range of motion for ankle joint for each woman. Transabdominal ultrasound: it will be used for measurement of Post-void residual volume PVR for each woman which is the volume of urine left in the bladder after micturition . Perineal ultrasound: it will be used to assess the posterior urethrovesical angle for each woman . X-ray radiography: lateral pelvic radiographs will be taken for each woman in order to objectify the individual pelvic tilt. Inclusion criteria include : Subjects will be postmenopausal women complaining from stress urinary incontinence Participants age will range from 60-70 years.Their BMI will not exceed 30 kg/m2. Exclusion criteria: previous history of cancer and radiotherapy, any disease that could interfere with the participation, lower urinary tract infections( Manshadi F. etal ) musculoskeletal problems; previous major abdominal or pelvic surgery; severe diseases; diabetes mellitus, a body mass index >30 kg/m2; intraureterine device implantation, pelvic organ prolapse and menopause (Cerruto M etal.)

ELIGIBILITY:
Inclusion Criteria:

Subjects will be 300 postmenopausal women suffering from stress urinary incontinence Participants age will range from 60-70 years.Their BMI will not exceed 30 kg/m2

Exclusion Criteria:

* previous history of cancer and radiotherapy, any disease that could interfere with the participation, lower urinary tract infections( Manshadi F. etal ) musculoskeletal problems; previous major abdominal or pelvic surgery; severe diseases; diabetes mellitus, a body mass index >30 kg/m2; intraureterine device implantation, pelvic organ prolapse and menopause (Cerruto M etal.)

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: 300 postmenopausal women suffering from stress urinary incontinence Participants age will range from 60-70 years.Their BMI will not exceed 30 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-29 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Post-void residual volume PVR | 30 minutes for every patient
  Transabdominal ultrasound
  it will be used for measurement of Post-void residual volume PVR for each woman which is the volume of urine left in the bladder after micturition
posterior urethrovesical angle | 30 minutes for every patient
  perineal ultrasound will be used to assesse the posterior urethrovesical angle for each woman
pelvic tilt | 30 minutes for every patient
  lateral pelvic radiographic xray will be taken for each woman in order to objectify the individual pelvic tilt

SECONDARY OUTCOMES:
ankle range of motion | 10 minutes for every patient
  goniometer will be used to measure the range of motion for ankle joint
BMI | 10 minutes for every patient
  weight height scale will be used to measure weight and height of each woman before starting this study